CLINICAL TRIAL: NCT04125615
Title: Resident Physician Burnout and Well-being: One Intervention and Its Impact
Brief Title: Resident Physician Burnout and Well-being
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 1612E02561
Record Dates: First submitted 2019-10-10; First posted 2019-10-14 (Actual); Last update posted 2019-10-14 (Actual); Status verified 2019-10

CONDITIONS: Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Protected Non-Clinical Time (Experimental): Protected non-clinical time
  Interventions: Behavioral: Protected Time Intervention
- Control Period (No Intervention): No protected non-clinical time

INTERVENTIONS:
Behavioral: Protected Time Intervention — Participants were assigned two hours of protected, non-clinical time by the chief resident of the service. Chief residents were instructed to assign this time when clinical learning opportunities were lowest. Each participant acted as their own control and was on the intervention phase of the study for the first or last 6 weeks of a quarterly rotation. Residents were concurrently assigned to the same phase of the study (intervention versus control). Participants were not specifically limited in what they could do during their non-clinical time, but they were encouraged to use this time in a way they felt would decrease their own personal burnout and increase their well-being, whether this be performing work-related administrative duties previously done on personal time or fulfilling obligations that are integral to personal health and well-being that can only be completed during normal business hours.
  Arms: Protected Non-Clinical Time

SUMMARY:
Pilot study shows that two hours of weekly protected non-clinical time is associated with decreased burnout and increased well-being in otolaryngology residents

DETAILED DESCRIPTION:
Burnout amongst physicians is high with resulting concern over quality of care. With burnout beginning early in training, much-needed data is lacking on interventions to decrease burnout and improve well-being amongst resident physicians. The primary objective was to design and evaluate the impact of a departmental-level burnout intervention for otolaryngology residents. The secondary objective was to describe how residents utilized and perceived the study intervention.

All current residents in the Department of Otolaryngology at the University of Minnesota were solicited for participation. Inclusion criteria included all residents willing to complete the study protocol. Exclusion criteria included the principal investigator. All 19 eligible residents consented to participate. All participants were assigned two hours of weekly, protected non-clinical time alternating with a control period of no intervention at 6 week intervals.

Burnout was measured by the Maslach Burnout Inventory (MBI) and Mini-Z Questionnaire (Mini-Z). Well-being was measured by the Resident and Fellow Well-Being Index (WBI) and a quality-of-life (QOL) single-item self-assessment (SA). In addition to baseline demographic survey, participants completed the aforementioned surveys at approximately 6-week intervals from October 2017 to July 2018.

ELIGIBILITY:
Inclusion Criteria:

- all resident physicians (PGY1 - PGY5) in the Department of Otolaryngology that were willing to complete the study protocol

Exclusion Criteria:

- principal investigator(s) were excluded from participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Maslach Burnout Inventory (MBI) Emotional Exhaustion (EE) Subscale | baseline, end of intervention (32 weeks)
  The MBI is a 22-item questionnaire with three subscales: emotional exhaustion (EE), depersonalization (DP), and personal achievement (PA). Lower EE and DP scores and higher PA are associated with decreased burnout. MBI subscale scores are calculated as the average of the component MBI items (9 items for MBI EE, 5 items for MBI DP, 8 items for MBI PA) with each scale resulting in MBI scale scores that ranged from 0 (Never) to 6 (Every day).
Change in Maslach Burnout Inventory (MBI) Depersonalization (DP) Subscale | baseline, end of intervention (32 weeks)
  The MBI is a 22-item questionnaire with three subscales: emotional exhaustion (EE), depersonalization (DP), and personal achievement (PA). Lower EE and DP scores and higher PA are associated with decreased burnout. MBI subscale scores are calculated as the average of the component MBI items (9 items for MBI EE, 5 items for MBI DP, 8 items for MBI PA) with each scale resulting in MBI scale scores that ranged from 0 (Never) to 6 (Every day).
Change in Maslach Burnout Inventory (MBI) Personal Achievement (PA) Subscale | baseline, end of intervention (32 weeks)
  The MBI is a 22-item questionnaire with three subscales: emotional exhaustion (EE), depersonalization (DP), and personal achievement (PA). Lower EE and DP scores and higher PA are associated with decreased burnout. MBI subscale scores are calculated as the average of the component MBI items (9 items for MBI EE, 5 items for MBI DP, 8 items for MBI PA) with each scale resulting in MBI scale scores that ranged from 0 (Never) to 6 (Every day).
Change in Mini-Z Questionnaire (Mini-Z) Question 3 | baseline, end of intervention (32 weeks)
  The Mini-Z is derived from the "Z" Clinician Questionnaire and has been validated with 10 stand-alone questions measuring feelings of burnout. For this study, only question 3 was used. This multiple-choice question assesses feelings of burnout using the participant's own definition. Answers range from A (I enjoy my work. I have no symptoms of burnout.) to E (I feel completely burned out. I am at the point where I may need to seek help.).
Change in Resident and Fellow Well-Being Index (WBI) | baseline, end of intervention (32 weeks)
  The WBI is a 7-item validated screening tool designed specifically for resident physicians to evaluate fatigue, depression, burnout, anxiety/stress, and mental/physical QOL. The WBI scale score is the total number of negative conditions that were experienced in the past month resulting in a scale score ranging from 0 - 7 with lower scores indicating higher well-being.
Change in Quality-of-Life (QOL) Single-Item Self-Assessment (SA) | baseline, end of intervention (32 weeks)
  The QOL SA has 5 response options to the question "Which of the following best describes your overall quality of life?" 0: As bad as it can be, 1: Somewhat bad, 2: Neutral, 3: Somewhat good, 4: As good as it can be, with higher QOL scores indicating higher quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Stevens, MD, Principal Investigator — University of Minenesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States